CLINICAL TRIAL: NCT04935749
Title: Epidemiologic Assessment of Diabetic Retinopathy in Egypt Using Ultrawide Field Fundus Photographs
Status: Recruiting | Type: Observational
Sponsor: Alexandria University (Other)
Collaborators: Joslin Diabetes Center (Other); Harvard Medical School (HMS and HSDM) (Other); I-care Ophthalmology Hospital (Unknown)
Responsible Party: Principal Investigator, Mohamed Ashraf Elmasry, Lecturer of Ophthalmology, Alexandria University
Other Study IDs: 0305153
Record Dates: First submitted 2021-05-29; First posted 2021-06-23 (Actual); Last update posted 2021-06-23 (Actual); Status verified 2021-06

CONDITIONS: Diabetic Retinopathy; Diabetic Macular Edema; Retinal Disease
Keywords: Ultra wide-field imaging; Diabetic retinopathy; Diabetes mellitus; Hand held cameras; Screening; Telemedicine; Artificial intelligence
MeSH Terms: conditions — Diabetic Retinopathy; Retinal Diseases; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Device: Ultra wide-field retinal imaging — Diabetic patients will be imaged with an ultra wide-field retinal imaging device (Optos, California). Patients will be imaged either with or without mydriasis.

SUMMARY:
In 2013, it was estimated that 16% (7.5 million) of all Egyptian adults between the ages of 20 and 79 years have type 2 diabetes and 2.6 million have diabetic retinopathy. A small pilot study looking at 323 patients with previously diagnosed diabetes mellitus (DM) and 183 patients with newly diagnosed DM found that the prevalence of diabetic retinopathy (DR) was 48.3% and 10.4% in each group respectively. By 2035, the Middle Eastern Region and Egypt is projected to have an over 96% increase in the diabetes population.

Ultrawide field (UWF) imaging is a novel technology that allows the visualization of approximately 82% of the retina in a single image. Its use in diabetic retinopathy (DR) has been widely explored both as a diagnostic as well as a screening tool. Using this technology, more of the peripheral retina can be readily visualized allowing significantly greater hemorrhages/microaneurysms, intraretinal microvascular abnormalities and non-perfusion to be detected. UWF imaging in patients with DM allowed the identification of a distinct sub-set of eyes with lesions that are predominantly distributed in the peripheral retina. Eyes with significantly greater DR lesions in the extended peripheral fields compared to their respective ETDRS fields are said to have predominantly peripheral lesions or PPL. Eyes with PPL are at greater risk of progressing to more advanced DR and developing proliferative diabetic retinopathy (PDR) after 4 years of follow up. The increased risk of vision threatening complications in eyes with PPL has made the identification of these eyes an essential part of DR evaluation and screening. Furthermore, the presence of lesions in the peripheral retina results in a more severe DR grade in approximately 20% of eyes thereby making this tool more accurate at grading DR severity. A recent DRCR retina network multicenter study established earlier findings confirming the validity of this tool in DR management.

I-care Ophthalmology Center will acquire the first UWF device in Egypt, the Optos California (Optos Plc, Dunfermline). Scanning laser ophthalmoscopy UWF imaging has been approved by both the FDA and EMA since 2011. Patients with DM, with or without known DR, will be imaged using the UWF imaging device both for diagnosis and screening purposes at I-care Ophthalmology center after informed consent. These images will be graded for the level of retinopathy and the presence/absence of PPL by certified trained graders. Internal validation and continuous quality control will routinely be conducted. Patients with vision threatening retinopathy (moderate non-proliferative diabetic retinopathy or worse, or the presence of diabetic macular edema) will be instructed to come back for further retinal evaluation and ancillary testing. Patients with mild retinopathy will be instructed to come for yearly follow up imaging. The expected duration for data collection will be 5-years, with interim data analysis on a yearly basis. The design although cross sectional, will have a prospective sub-analysis group in patients who have repeat imaging.

Data collection and imaging will be conducted in Egypt and anonymized deidentified data will be shared with the Joslin Diabetes Center, Harvard Ophthalmology Department for joint research purposes. Data will be analyzed for the prevalence of DR and the distribution of DR severity levels in the studied population. In addition, the presence and absence of PPL and its association with DR progression will be studied. Non-modifiable (duration of DM, age of onset, type of DM etc.) and modifiable risk factors (HbA1c, hypertension, hyperlipidemia etc.) for increased risk of DR progression will also be analyzed. Sensitivity analysis will explore the sensitivity/specificity of initial DR grading compared to trained retina specialists.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus

Exclusion Criteria:

* Patients unable or unwilling to be imaged

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with diabetes who present for imaging as part of a local diabetic retinopathy screening program (DRSP) will be imaged using an ultrawide field camera.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2021-07-01 (Estimated); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Epidemiology | 1 year
  Describing the distribution of different DR severity levels using UWF imaging
DR Progression | 4 years
  Assessing the number of patients with at least 4 years of follow up who have a 2 step or more DR progression
Progression to PDR | 4 years
  Assessing the number of patients with at least 4 years of follow up who progress to PDR
Epidemiology | 1 year
  Prevalence of predominantly peripheral lesions (PPL) in eyes with DR using UWF imaging

CONTACTS AND LOCATIONS:
Locations (1):
- I-care Ophthalmology Center, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No